CLINICAL TRIAL: NCT05823883
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed Dose Combination of DW6014 and Loose Combination of Each Component in Healthy Adult Volunteers in Fed Condition
Brief Title: This Study is to Compare and Evaluate the Safety and Pharmacokinetic Characteristics (PK) After Administration of DW6014 and Each Component in Healthy Adult Volunteers in Fed Condition.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW6014-I-2
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: DW6014
MeSH Terms: interventions — empagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Empagliflozin and Metformin Period 2: DW6014
  Interventions: Drug: DW6014
- Sequence B (Experimental): Period 1: DW6014 Period 2: Empagliflozin and Metformin
  Interventions: Drug: DW6014

INTERVENTIONS:
Drug: DW6014 — Drug: DW6014 Single oral administration of DW6014 in fed condition
  Drug: Empagliflozin and Metformin Combination oral administration of Empagliflozin and Metformin in fed condition
  Other Names: Empagliflozin and Metformin

SUMMARY:
This study is to compare and evaluate the safety and pharmacokinetic characteristics (PK) after administration of DW6014 and each component in healthy adult volunteers in fed condition.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, Oral, Single-dose, two-way crossover study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged up to 19 years
* Subjects weighing at least 50.0 kg with a BMI between 18.0 kg/m2 and 30.0 kg/m2
* Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
* Subjects considered eligible for the study participation in accordance to the results of clinical laboratory tests, vital signs, physical examinations and 12-lead ECG conducted at the time of screening, based on the investigational product (IP) characteristics
* Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

* Subjects with any clinically significant hepatic, renal, nervous, respiratory, endocrine, circulatory, tumor, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases or other medical history
* Subject with galactose intolerance, Lapp lactase deficience, glucose-galactose malabsorption or other genetic problem
* Subject following gastrointestinal diseases or gastrointestinal surgery that may affect the absorption of the IP
* Pregnant subjects with a positive urine HCG(human chorionic gonadotropin) test, or lactating female subjects
* Subject with a medical history of hypersensitivity reactions (anaphylaxis or antibiotics etc.) to containing empagliflozin and metformin components, formulation additives, and other drugs (aspirin, antibiotics, biguanide drugs, etc.) or clinically significant hypersensitivity reactions
* Subjects with clinically significant 12-lead ECG findings at the time of screening
* Subjects with a past history of drug abuse or a positive urine drug test
* Subjects with SBP(systolic blood pressure) ≥ 150 mmHg or ≤ 90 mmHg; DBP(diastolic blood pressure) ≥ 100 mmHg or ≤ 60 mmHg; Pulse Rate ≤ 40 bpm or ≥ 100 bpm at the time of screening
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects who have administered any prescription drugs or herbal medicines that may affect the characteristics of clinical investigational drugs within 2 weeks prior to the first administration date, or have administered any over-the-counter (OTC) or vitamin preparations within 10 days
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration Before the first administration date whole blood donation within 2 months or component blood donation within 1 month or received a blood transfusion within 1 month, or the subject who cannot forbid transfusion from the time of obtaining ICF(informed consent form) until PSV(post-study visit)
* Subjects who have consistently drunk alcohol within 6 months
* Subjects who have smoked more than 10 cigarettes/day on average
* Subjects who have eaten or cannot refrain from eating grapefruit (grapefruit)-containing food from 48 hours before the first administration until the time of PSV(post-study visit)
* Subjects who have consumed or cannot refrain from consuming caffeine-containing food during the period from 24 hours prior to administration of each period to the time of the last blood sampling
* Subjects who have done and are unable to refrain from strenuous activity
* Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception
* Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | 48 hour
  AUC0-t of Metformin
Cmax | 48 hour
  Cmax of Metformin

SECONDARY OUTCOMES:
Tmax | 48 hour
  Tmax of Metformin
AUCinf | 48 hour
  AUCinf of Metformin
t1/2 | 48 hour
  t1/2 of Metformin
CL/F | 48 hour
  CL/F of Metformin
Vd/F | 48 hour
  Vd/F of Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea